CLINICAL TRIAL: NCT04114929
Title: Is a Threshold Based Model a Superior Method at Improving Cardiorespiratory Fitness in Patients Attending Phase IV Cardiac Rehabilitation
Brief Title: Is Threshold-based Training Superior in Cardiac Rehabilitation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19
Sponsor: University of Central Lancashire (Other)
Collaborators: University of Hull (Other); Leeds Beckett University (Other); Sheffield Hallam University (Other)
Responsible Party: Principal Investigator, Stefan Birkett, Lecturer In Exercise Science, University of Central Lancashire
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UCentalLancashire
Record Dates: First submitted 2019-09-28; First posted 2019-10-03 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: Cardiac Rehabilitation
Keywords: ventilatory anaerobic threshold; Intensity; Exercise Dose; Standard care
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Patients will randomised either to threshold-based training or standard care
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Threshold-Based (Experimental): Patients will be prescribed exercise based on ventilatory thresholds from a maximal cardiopulmonary exercise test
  Interventions: Other: Threshold-based Training
- Standard Care (Active Comparator): Patients will be prescribed exercise based on standard guidelines
  Interventions: Other: Standard Care

INTERVENTIONS:
Other: Threshold-based Training — Specific ventilatory markers determined from a cardiopulmonary test and the correlating heart rate will be used to determine exercise intensity
  Arms: Threshold-Based
Other: Standard Care — Using the standard care cardiac rehabilitation guidelines exercise will be based on estimated heart rate maximum followed by the karvonan method to calculate 40-70% heart rate reserve
  Arms: Standard Care

SUMMARY:
This study evaluates two methods of prescribing exercise intensity in a Phase IV cardiac rehabilitation programme. One method is using specific ventilatory markers and the other following standard care guidelines.

DETAILED DESCRIPTION:
Coronary heart disease (CHD) is one of the United Kingdom's (UK) biggest killers. In the UK alone 175,000 myocardial infarctions are recorded annually. While these numbers are significant advances in preventative therapy and medical treatment have contributed to an overall reduction in mortality in the UK. As such there is a growing need for effective secondary prevention. To lower the financial burden on the National Health Service (NHS), cardiac rehabilitation (CR) facilitates a systematic and multidisciplinary approach to secondary prevention aimed to improve functional capacity and health-related quality of life, lower rehospitalisation rates and reduce all-cause and cardiovascular mortality with exercise training being the cornerstones.

A 2016 Cochrane review found benefits of exercise-based CR for patients with coronary artery disease. Both cardiovascular mortality and hospital readmissions were reduced, when compared with a no-exercise control. However, in contrast to previous systematic reviews and meta-analyses, there was no significant reduction in risk of reinfarction or all-cause mortality. Further a recent systematic review and meta-analysis (2018) found no differences in outcomes between exercise-based CR and a no-exercise control at their longest follow-up period for: all-cause mortality or cardiovascular mortality. The authors also found a small reduction in hospital admissions of borderline statistical significance. One possible answer to the above findings is the under dosage of exercise intensity and duration in UK CR. A recent multicentre study of routine UK-based CR (current clinical practice) indicated that the 'exercise dose' within outpatient UK CR may be insufficient to meaningfully improve cardiorespiratory fitness (CRF) when compared with international programmes. Given the prognostic relevance of improving CRF and that exercise and physical activity has a 'dose-response' relationship with cardiovascular disease risk, these findings may explain why UK CR programmes do not appear to improve patient survival.

UK-based guidelines advocate a percentage range-based method for prescribing exercise intensity. However, there are a number of limitations of this method. The investigators and others have recently shown that prescribing exercise intensity using percentage heart rate reserve (%HRR) can lead to patients receiving different exercise training doses from what would be historically viewed as the same exercise training intervention. Prescribing exercise based on %HRR ignores the important role that metabolic perturbations play in stimulating physiological adaptation in response to exercise training. The ventilatory anaerobic threshold (VAT) is an important objective metabolic threshold that indicates when incrementally greater contributions from anaerobic metabolism are required to sustain further increases in workload. The VAT has been proposed as a minimum exercise training intensity that must be exceeded in order to improve aerobic fitness. Compelling data has shown that the occurrence of the VAT is patient-specific, and can occur at different percentage of a patient's HRR. Basing an exercise training programme on estimated, or even directly measured %HRR could therefore result in heart rate training zones being set either above, or below the VAT. Patients who are prescribed the 'same' exercise training programme based on %HRR could be exposed to different metabolic stimuli and therefore a different exercise training dose. This may explain why some patients appear to 'respond' to a treatment, whilst others may be classified as "non-responders." Prescribing exercise that can improve CRF for patients attending CR is essential, and greater consideration for how exercise is prescribed in a community-based setting is required.

Given the VAT is a significant threshold, with evidence reporting it to be a superior method, comparisons to the %HRR method are limited in clinical populations. As such the primary focus of the study is to compare the effectiveness of a threshold-based model (ventilatory threshold) versus a relative percent model (%HRR) for improving cardiorespiratory fitness in patient attending Phase IV community based cardiac rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Patient has read and understood the Patient Information Sheet
* Diagnosis of coronary heart disease (CHD) including myocardial infarction(MI), coronary artery bypass graft (CABG) surgery, elective percutaneous coronary intervention (PCI) or exertional angina.

  . Diagnosis of heart failure
* Aged between 18 and 85 years
* Absence of contraindications to exercise testing and training
* Clinically stable (symptoms and medication)
* Patient is able to and has given written informed consent
* Able to comply with guidelines for participation in exercise testing & prescription

Exclusion Criteria:

• Clinically Unstable

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2021-11-01 (Estimated); Study Completion 2022-08-01 (Estimated)

PRIMARY OUTCOMES:
Peak Oxygen Consumption Change | Baseline & 3 months
  Peak Oxygen Consumption as determined by a cardiopulmonary exercise test

SECONDARY OUTCOMES:
Health Related Quality of Life Change (EuroQoL EQ-5D) | Baseline & 3 months
  Quality of Life as determined by the Health Related Quality of Life Questionnaire. The questionnaire five sections, mobility, self-care, usual activities, pain/discomfort and anxiety and depression. The scoring system is not displayed on the questionnaire however when evaluating runs in order of severity (0-4). A 0-100 scale follows where a patient will score their health status. 100 means the best health they can imagine and 0 means the worst

CONTACTS AND LOCATIONS:
Locations (1):
- School of Sport and and Health Sciences, Preston, United Kingdom